CLINICAL TRIAL: NCT04731558
Title: Pre- Vs Postoperative Thromboprophylaxis for Liver Resection - a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Pre- Vs Postoperative Thromboprophylaxis for Liver Resection
Acronym: PREPOSTEROUS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Academy of Finland (Other); The Finnish Medical Association (Other)
Responsible Party: Principal Investigator, Ville Sallinen, Principal investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HYKS-PREPOSTEROUS
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Liver Cancer; Surgery; Thrombosis, Deep Vein; Embolism, Pulmonary; Bleeding
MeSH Terms: conditions — Liver Neoplasms; Venous Thrombosis; Pulmonary Embolism; Hemorrhage | interventions — Enoxaparin; Tinzaparin; Dalteparin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative thromboprophylaxis (Experimental): Preoperatively initiated tromboprophylaxis
  Interventions: Drug: enoxaparin or tinzaparin or dalteparin
- Postoperative thromboprophylaxis (Other): Postoperatively initiated thromboprophylaxis
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: enoxaparin or tinzaparin or dalteparin — Thromboprophylaxis initiated approximately 14 hours prior to the planned liver resection skin incision. Thromboprophylaxis can be initiated using enoxaparin (20 - 40 mg), tinzaparin (2500 - 4500 IU), or dalteparin (2500 - 5000 IU), with the dose based on patient's renal function
  Arms: Preoperative thromboprophylaxis
Drug: No intervention — No preoperative thromboprophylaxis.
  Arms: Postoperative thromboprophylaxis

SUMMARY:
Thromboprophylaxis for liver surgery can be commenced either preoperatively or postoperatively. Despite a clear trade-off between thrombosis and bleeding in liver surgery patients, there is no international consensus when thrombosis prophylaxis should be commenced in patients undergoing liver surgery. As far as we know, there are no prospective randomized trials in this field, and current guidelines are unfortunately based on very low quality evidence, that is, a few retrospective studies and expert opinion. Both American and European thromboprophylaxis guidelines for abdominal cancer surgery support the preoperative initiation of thromboprophylaxis, but these guidelines do not specifically address the increased bleeding risk associated with liver surgery. On the contrary, Dutch guidelines recommend postoperative thromboprophylaxis only, because of lack of evidence for preoperative thromboprophylaxis. Traditionally, many liver surgery units have been reluctant in using preoperative thromboprophylaxis due to the potentially increased risk of bleeding complications. Enhanced Recovery After Surgery (ERAS) Society Guidelines recommend preoperative thromboprophylaxis in liver surgery, but the guidelines provide no supporting evidence for this recommendation. Overall, the amount of evidence is scarce and somewhat contradictory in this clinically relevant field of thromboprophylaxis in liver surgery. The aim of this study is to compare pre- and postoperatively initiated thromboprophylaxis regimens in liver surgery in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing liver resection

Exclusion Criteria:

* Patient on anticoagulative medication (heparin, low-molecular weight heparin, warfarin, direct oral anticoagulants) during last month pre-surgery
* Emergency operation (e.g. for trauma or infection)
* Age < 18 years
* Allergy or other contraindication to planned low-molecular weight heparin
* Inability to give written informed consent
* Liver resection not performed (removed from analyses after randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolisms | within 30 days from liver resection
  Number of patients with venous thromboembolism defined as either 1) symptomatic deep venous thromboembolism (includes all deep veins e.g. all extremities, portal vein, and superior mesenteric) diagnosed using ultrasound or computed tomography or magnetic resonance imaging, or in re-laparatomy/surgery, 2) pulmonary embolism diagnosed using computed tomography, magnetic resonance imaging, or lung perfusion imaging, or 3) death due to venous thromboembolism

SECONDARY OUTCOMES:
Posthepatectomy haemorrhage | within 30 days from liver resection
  Number of patients with posthepatectomy haemorrhage, any grade in ISGLS classification
Postoperative complications | within 30 days from liver resection
  Comprehensive Complication Index - score
Length of postoperative hospital stay | within 30 days from liver resection
  Length of postoperative hospital stay, days
Blood transfusion | during and within 30 days from liver resection
  Total amount of transfused red blood cells, units

CONTACTS AND LOCATIONS:
Locations (7):
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Norway (2):
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: Undecided